CLINICAL TRIAL: NCT03283761
Title: A Phase II Study of FOLFOX Combined With Nab-Paclitaxel (FOLFOX-A) in the Treatment of Metastatic or Advanced Unresectable Gastric, Gastro-Esophageal Junction Adenocarcinoma. Big Ten Cancer Research Consortium: BTCRC-GI15-015
Brief Title: FOLFOX-A in the Treatment of Metastatic or Advanced Unresectable Gastric, Gastro-Esophageal Junction Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Al B. Benson, III, MD (Other)
Collaborators: Celgene Corporation (Industry); Big Ten Cancer Research Consortium (Other)
Responsible Party: Sponsor-Investigator, Al B. Benson, III, MD, Sponsor-Investigator, Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC-GI15-015
Record Dates: First submitted 2017-09-13; First posted 2017-09-14 (Actual); Results first posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Gastro-Esophageal Junction Adenocarcinoma; Gastric Cancer
Keywords: FOLFOX; Nab-Paclitaxel
MeSH Terms: conditions — Stomach Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Masking Description: Open-Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): All patients in Stage I (N=12) and Stage II (N=25) will receive FOLFOX-A on days 1 and 15 of each cycle (1 cycle = 28 days). Nab-paclitaxel will be given at a dose of 150 mg/m^2 IV over 30 minutes, followed by oxaliplatin IV 85 mg/m^2 and leucovorin IV 400 mg/m^2 over 2 hours, and 5-FU as a continuous IV infusion over Day 1 and Day 2 (for a total dose of 2400mg/m^2 over 46-48 hours.). Radiographic assessment will be performed at baseline and every other cycle (starting with Cycle 3) to evaluate response to treatment by RECIST Version 1.1 guidelines. Patients may continue to receive treatment until disease progression or unacceptable toxicity.
  Interventions: Drug: Nab-paclitaxel 150 mg/m^2; Drug: Oxaliplatin 85 mg/m^2; Drug: 5-FU 1200 mg/m^2 x 2 D; Drug: Leucovorin 400 mg/m^2

INTERVENTIONS:
Drug: Nab-paclitaxel 150 mg/m^2 — Stage I (N=12), on day 1 and day 15 Stage II (N= 25), on day 1 and day 15
  Other Names: Abraxane®
Drug: Oxaliplatin 85 mg/m^2 — Stage I (N= 12), on day 1 and day 15 Stage II (N= 25), on day 1 and day 15
  Other Names: Eloxatin
Drug: 5-FU 1200 mg/m^2 x 2 D — Stage I (N= 12), on day 1 and day 15-16 Stage II (N= 25),on day 1 and day 15-16
  Other Names: Adrucil; Fluorouracil
Drug: Leucovorin 400 mg/m^2 — Stage I (N= 12),on day 1 and day 15 Stage II (N= 25), on day 1 and day 15

SUMMARY:
This is an open label, single-arm phase II, multi-institutional trial to evaluate the efficacy and safety of the combination of nab-paclitaxel and FOLFOX (FOLFOX-A) as first line therapy for patients diagnosed with histologically-confirmed advanced gastric/GEJ adenocarcinoma.

DETAILED DESCRIPTION:
All patients will receive FOLFOX-A on days 1 and 15 of each cycle (1 cycle = 28 days). Nab-paclitaxel will be given at a dose of 150 mg/m2 IV over 30 minutes, followed by oxaliplatin IV 85 mg/m2 and leucovorin IV 400 mg/m2 over 2 hours, and 5-FU as a continuous IV infusion over Day 1 and Day 2 (for a total dose of 2400mg/m2 over 46-48 hours.). Radiographic assessment will be performed at baseline and every other cycle (starting with Cycle 3) to evaluate response to treatment by RECIST Version 1.1 guidelines. Patients may continue to receive treatment until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following applicable inclusion criteria to participate in this study:

* Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of 0-1 within 28 days prior to registration.
* Histologically-confirmed advanced or metastatic unresectable gastric carcinoma, or adenocarcinoma of the gastroesophageal junction.
* Prior neoadjuvant or adjuvant chemotherapy, hormonal therapy, immunotherapy, radiation or chemoradiotherapy must have been completed at least 6 months prior to documented recurrence or metastatic disease. NOTE: patients must not have received previous systemic treatment for metastatic disease.
* Evaluable disease according to RECIST v1.1 for solid tumors, within 28 days prior to registration.
* Demonstrate adequate organ function as described below; all screening labs to be obtained within 28 days prior to registration.

  * Bilirubin < 1.5 mg/dL
  * Patients must have adequate liver function: AST and ALT < 2.5 x upper limit of normal, alkaline phosphatase < 2.5 x upper limit of normal, unless bone or liver metastasis is present (≤5 x upper limit of normal).
  * Patients must have adequate bone marrow function: Platelets >100,000 cells/mm3 (transfusion independent, defined as not receiving platelet transfusions within 7 days prior to laboratory sample), Hemoglobin > 9.0g/dL and ANC > 1,500 cells/mm3.
  * Patients must have adequate renal function: creatinine <1.5 mg/dL or creatinine clearance ≥60mL/min is recommended; however, institutional norms are acceptable.
* Females of child-bearing potential (defined as a sexually mature woman who (1) has not undergone hysterectomy [the surgical removal of the uterus] or bilateral oophorectomy [the surgical removal of both ovaries] or (2) has not been naturally postmenopausal for at least 24 consecutive months [i.e., has had menses at any time during the preceding 24 consecutive months]) must:

  * Either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis), or agree to use and be able to comply with effective contraception without interruption 28 days prior to starting investigational product (IP), and while on study medication (including dose interruptions) and for 30 days following the last dose of IP; and
  * Have a negative serum pregnancy test (β -hCG) result at screening and agree to ongoing pregnancy testing prior to each treatment and after the end of study therapy. This applies even if the subject practices true abstinence* from heterosexual contact.
  * Male subjects must practice true abstinence* or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for 6 months following IP discontinuation, even if he has undergone a successful vasectomy.

    * NOTE: True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception].

Exclusion Criteria

Subjects meeting any of the criteria below may not participate in the study:

* Her-2 positive gastric tumor.
* Treatment with any investigational products within 28 days prior to study registration.
* Preexisting peripheral neuropathy is not allowed from any cause.
* Known history of Human Immunodeficiency Virus (HIV) or Hepatitis C (baseline testing is not required).
* Patients with active sepsis or pneumonitis
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to trial registration and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial registration.
* Known hypersensitivity to fluorouracil (5-FU), oxaliplatin, or other platinum agents.
* Known hypersensitivity to nab-paclitaxel or any of its excipients.
* History of slowly progressive dyspnea and unproductive cough, or pulmonary conditions such as sarcoidosis, silicosis, idiopathic pulmonary fibrosis, hypersensitivity pneumonitis or multiple allergies. See section 6.5.1.
* Has known dihydropyrimidine dehydrogenase deficiency (DPD) deficiency (testing not required)
* Ongoing or active infection requiring systemic treatment (must be afebrile for ≥ 48 hours prior to study registration)
* Uncontrolled intercurrent illness including, but not limited to any of the following:

  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
* Known additional malignancy within the past 3 years. Exceptions include treated localized basal cell or squamous cell carcinoma of the skin, in situ cervical or vulvar carcinoma that has undergone potentially curative therapy, superficial bladder tumors (Ta, Tis & T1), ductal carcinoma in situ (DCIS) of the breast and low grade prostate cancer (Gleason sore 6). Any cancer curatively treated > 3 years prior to registration with no clinical evidence of recurrence is permitted.
* Psychiatric illness/social situations that would limit compliance with study requirements.
* Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2023-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Al B. Benson, MD, Principal Investigator — Big Ten Cancer Research Consortium
Locations (8):
- United States (8):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Univeristy of Illinois Cancer Center, Chicago, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Michigan State University, Lansing, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Big Ten Cancer Research Consortium Website — http://www.bigtencrc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Nab-paclitaxel and FOLFOX-A: All patients in Stage I (N=12) and Stage II (N=25) will receive FOLFOX-A on days 1 and 15 of each cycle (1 cycle = 28 days). Nab-paclitaxel will be given at a dose of 150 mg/m^2 IV over 30 minutes, followed by oxaliplatin IV 85 mg/m^2 and leucovorin IV 400 mg/m^2 over 2 hours, and 5-FU as a continuous IV infusion over Day 1 and Day 2 (for a total dose of 2400mg/m^2 over 46-48 hours.). Radiographic assessment will be performed at baseline and every other cycle (starting with Cycle 3) to evaluate response to treatment by RECIST Version 1.1 guidelines. Patients may continue to receive treatment until disease progression or unacceptable toxicity.
  Nab-paclitaxel 150 mg/m^2: Stage I (N=12), on day 1 and day 15 Stage II (N= 25), on day 1 and day 15
  Oxaliplatin 85 mg/m^2: Stage I (N= 12), on day 1 and day 15 Stage II (N= 25), on day 1 and day 15
  5-FU 1200 mg/m^2 x 2 D: Stage I (N= 12), on day 1 and day 15-16 Stage II (N= 25),on day 1 and day 15-16
  Leucovorin 400 mg/m^2: Stage I (N= 12),on day 1 and day 15 Stage II (N= 25), on day 1 and day 15
Period: Study Treatment
Arm/Group | Nab-paclitaxel and FOLFOX-A
Started | 39
Completed | 0
Not Completed | 39
Not completed — Patient Non-Compliance | 1
Not completed — Alternative Cancer Therapy | 7
Not completed — Disease progression | 21
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 4
Not completed — Pre-existing GI bleed and chronic anemia from that led to hospitalization and going off trial. | 1
Not completed — Symptomatic Deterioration | 1
Not completed — Screen Failure Before Therapy Start | 1
Period: Follow up
Arm/Group | Nab-paclitaxel and FOLFOX-A
Started | 38 (Treatment and Follow up both are at different time period. Therefore, the number of subjects to start follow up is not equal to the number of subjects who have completed treatment.)
Completed | 0
Not Completed | 38
Not completed — Lost to Follow-up | 1
Not completed — Symptomatic Deterioration | 1
Not completed — Death | 29
Not completed — study terminated | 4
Not completed — Primary Investigator Withdrawal | 1
Not completed — Switched to alternative therapy | 1
Not completed — Subject is now in Hospice | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nab-paclitaxel and FOLFOX-A
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 63 [20 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 34
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Fairview Southdale Cancer Clinic | 1
  United States: M Health Fairview Clinics and Surgery Center | 2
  United States: Northwestern Memorial Hospital | 20
  United States: Rutgers Cancer Institute of New Jersey | 2
  United States: University of Illinois Hospital and Health Systems (Outpatient Cancer Center) | 2
  United States: University of Iowa Hospitals and Clinics | 7
  United States: University of Wisconsin Clinical Science Center | 5
ECOG [Count of Participants; unit: Participants] — Performance status Definition 0 Fully active; no performance restrictions.
  1. Strenuous physical activity restricted; fully ambulatory and able to carry out light work.
  2. Capable of all self-care but unable to carry out any work activities. Up and about >50% of waking hours.
  3. Capable of only limited self-care; confined to bed or chair >50% of waking hours.
  4. Completely disabled; cannot carry out any self-care; totally confined to bed or chair.
  Participants
    0 | 20
    1 | 19
T Stage [Count of Participants; unit: Participants] — TX: no information about the primary tumor, or it can't be measured;T (T3,T4) The higher the T number, the larger the tumor and/or the more it has grown into nearby tissues;NX: no information about the nearby lymph nodes, or they can't be assessed;N0:nearby lymph nodes do not contain cancer;N (N1, N2,N3) might describe the size, location, and/or the number of nearby lymph nodes affected by cancer. The higher the N number, the greater the cancer spread to nearby lymph nodes;M0:no distant cancer spread has been found;M1:cancer has been found to have spread to distant organs or tissues.
  Participants
    T3 | 13
    T4 | 5
    TX | 19
    Unknown T stage | 2
    N0 | 4
    N1 | 4
    N2 | 6
    N3 | 3
    NX | 20
    Unknown N stage | 2
    M0 | 2
    M1 | 35
    Unknown M stage | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective response rate will be calculated by combining the number of subjects who achieve complete response and partial response per RECIST 1.1 criteria.Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Complete response is defined as disappearance of all target lesions. Any pathological lymph nodes(whether target or non-target) must have reduction in short axis to <10 mm.
Time Frame: From C1D1 until death or up to a maximum of 36 months
Population: 35 subjects out of 39 enrolled subjects were evaluable for objective response.
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-paclitaxel and FOLFOX-A
Number analyzed (Participants) | 35
Participants | 15

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined by the date of the start of treatment to date of death from any cause.
Time Frame: From C1D1 until death or up to a maximum of 52 months
Population: one subject out of 39 enrolled subject was a screen failure before start of therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-paclitaxel and FOLFOX-A
Number analyzed (Participants) | 38
months | 10.6 [8.8 to 20.7]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression free survival is defined as the time of treatment initiation until the criteria for disease progression per RECIST1.1 are met or until the date of a death event (any cause). Progressive disease is defined as at least a 20% increase in the sum of the diameters of target lesions,taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: From C1D1 until death or up to a maximum of 36 months
Population: one subject out of 39 enrolled subject was a screen failure before start of therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-paclitaxel and FOLFOX-A
Number analyzed (Participants) | 38
months | 6.6 [5.7 to 12.9]

4. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression is defined as the time from registration date until the criteria for disease progression per RECIST1.1 are met. Progressive disease is defined as at least a 20% increase in the sum of the diameters of target lesions,taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: From C1D1 until PD or up to a maximum of 36 months
Population: one subject out of 39 enrolled subject was a screen failure before start of therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nab-paclitaxel and FOLFOX-A
Number analyzed (Participants) | 38
months | 11.26 [5.68 to 26.65]

5. Secondary Outcome: Number of Subjects Achieve Best Overall Response of CR, PR, SD and PD
Description: Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Complete response is defined as disappearance of all target lesions. Any pathological lymph nodes(whether target or non-target) must have reduction in short axis to <10 mm. Stable disease is defined as neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study. Progressive disease is defined as at least a 20% increase in the sum of the diameters of target lesions,taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: From C1D1 until PD or up to a maximum of 36 months
Population: one subject out of 39 enrolled subject was a screen failure before start of therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-paclitaxel and FOLFOX-A
Number analyzed (Participants) | 38
Participants
  Number of subjects with Complete Response as best RECIST response | 1
  Number of subjects with Partial Response as best RECIST response | 14
  Number of subjects with Stable Disease as best RECIST response | 13
  Number of subjects with Progressive Disease as best RECIST response | 7
  Number of subjects with no responses recorded | 3

6. Secondary Outcome: Disease Control Rate (DCR)
Description: The disease control rate is the proportion of all subjects with stable disease (SD) , or partial response (PR), or complete response (CR) according to RECIST 1.1, from the start of treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the start of treatment). Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Complete response is defined as disappearance of all target lesions. Any pathological lymph nodes(whether target or non-target) must have reduction in short axis to <10 mm. Stable disease is defined neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: From C1D1 until PD or up to a maximum of 36 months
Population: 35 subjects out of 39 enrolled subjects were evaluable for response.
Measure: Number; unit: percentage of participants
Arm/Group | Nab-paclitaxel and FOLFOX-A
Number analyzed (Participants) | 35
percentage of participants | 80

7. Secondary Outcome: Safety and Toxicity Profile of the Combination of Nab-paclitaxel and FOLFOX
Description: Safety and tolerability of abemaciclib in the combination of nab-paclitaxel and FOLFOX in patients with metastatic or advanced unresectable gastric, gastro-esophageal junction adenocarcinoma., assessed by NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.
Time Frame: From C1D1 until death or up to a maximum of 52 months
Population: one subject out of 39 enrolled subject was a screen failure before start of therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-paclitaxel and FOLFOX-A
Number analyzed (Participants) | 38
Participants
  Number of patients had at least one adverse event of any toxicity grade | 38
  Number of patients had at least one toxicity of grade 3 or greater adverse event | 32
  Number of patients had at least one grade 3 or greater treatment related adverse event | 32
  Number of patients having serious adverse event | 21

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from week 1 of treatment and every chemotherapy cycles thereafter, for up to 52 months or until unacceptable toxicity. All-Cause Mortality was assessed from week 1 of treatment and every chemotherapy cycles thereafter, for up to 52 months or until unacceptable toxicity
Description: An Adverse Event is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Arm/Group | Nab-paclitaxel and FOLFOX-A
All-Cause Mortality (participants affected / at risk) | 29/38
Serious Adverse Events (participants affected / at risk) | 22/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nab-paclitaxel and FOLFOX-A (N=38)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2)
ANEMIA (Blood and lymphatic system disorders) | 3 (3)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1)
BRONCHIAL INFECTION (Infections and infestations) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (2)
DEPRESSION (Psychiatric disorders) | 1 (2)
DIARRHEA (Gastrointestinal disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1)
ENCEPHALOPATHY (Nervous system disorders) | 2 (3)
GASTRIC HEMORRHAGE (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 1 (3)
LOWER GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1)
LUNG INFECTION (Infections and infestations) | 1 (1)
MULTI-ORGAN FAILURE (General disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 2 (2)
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 2 (2)
PAIN (General disorders) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1)
PERICARDITIS (Cardiac disorders) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (1)
SEPSIS (Infections and infestations) | 2 (2)
SKIN INFECTION (Infections and infestations) | 1 (1)
STROKE (Nervous system disorders) | 1 (1)
UPPER GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 2 (2)
VERTIGO (Ear and labyrinth disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nab-paclitaxel and FOLFOX-A (N=38)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 15 (27)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1)
AKATHISIA (Nervous system disorders) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 8 (21)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 9 (28)
ALLERGIC REACTION (Immune system disorders) | 1 (2)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 6 (6)
ALOPECIA (Skin and subcutaneous tissue disorders) | 16 (18)
AMNESIA (Nervous system disorders) | 1 (1)
ANEMIA (Blood and lymphatic system disorders) | 24 (67)
ANOREXIA (Metabolism and nutrition disorders) | 23 (39)
ANXIETY (Psychiatric disorders) | 14 (17)
AORTIC VALVE DISEASE (Cardiac disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (3)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 6 (6)
ASCITES (Gastrointestinal disorders) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 8 (15)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 8 (8)
BLOATING (Gastrointestinal disorders) | 6 (7)
BLOOD AND LYMPHATIC SYSTEM DISORDERS - OTHER, SPECIFY (Blood and lymphatic system disorders) | 4 (27)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1)
BLURRED VISION (Eye disorders) | 3 (4)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 4 (5)
BRUISING (Injury, poisoning and procedural complications) | 3 (3)
BUTTOCK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
CARDIAC DISORDERS - OTHER, SPECIFY (Cardiac disorders) | 5 (6)
CATHETER RELATED INFECTION (Infections and infestations) | 1 (1)
CHEST PAIN - CARDIAC (Cardiac disorders) | 1 (2)
CHILLS (General disorders) | 5 (6)
CHOLESTEROL HIGH (Investigations) | 5 (5)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1 (1)
COGNITIVE DISTURBANCE (Nervous system disorders) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1)
CONCENTRATION IMPAIRMENT (Nervous system disorders) | 2 (2)
CONFUSION (Psychiatric disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 28 (44)
COUGH (Respiratory, thoracic and mediastinal disorders) | 11 (13)
CREATININE INCREASED (Investigations) | 3 (3)
DEHYDRATION (Metabolism and nutrition disorders) | 8 (11)
DELIRIUM (Psychiatric disorders) | 1 (1)
DENTAL CARIES (Gastrointestinal disorders) | 1 (1)
DEPRESSION (Psychiatric disorders) | 5 (8)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (2)
DIARRHEA (Gastrointestinal disorders) | 25 (50)
DIZZINESS (Nervous system disorders) | 11 (12)
DRY MOUTH (Gastrointestinal disorders) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 (3)
DYSARTHRIA (Nervous system disorders) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 11 (13)
DYSPEPSIA (Gastrointestinal disorders) | 16 (18)
DYSPHAGIA (Gastrointestinal disorders) | 18 (24)
DYSPHASIA (Nervous system disorders) | 3 (3)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 5 (8)
EAR AND LABYRINTH DISORDERS - OTHER, SPECIFY (Ear and labyrinth disorders) | 2 (3)
EAR PAIN (Ear and labyrinth disorders) | 1 (1)
EDEMA LIMBS (General disorders) | 12 (13)
ENDOCARDITIS INFECTIVE (Infections and infestations) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 5 (5)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 2 (2)
ERYTHRODERMA (Skin and subcutaneous tissue disorders) | 1 (1)
EXTRAPYRAMIDAL DISORDER (Nervous system disorders) | 1 (1)
EYE DISORDERS - OTHER, SPECIFY (Eye disorders) | 1 (1)
FACIAL PAIN (General disorders) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 5 (8)
FATIGUE (General disorders) | 32 (63)
FEVER (General disorders) | 11 (12)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3)
FLU LIKE SYMPTOMS (General disorders) | 3 (5)
FLUSHING (Vascular disorders) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 2 (3)
GASTRITIS (Gastrointestinal disorders) | 1 (1)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 16 (17)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 11 (15)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 1 (1)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (General disorders) | 2 (10)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 5 (6)
GINGIVAL PAIN (Gastrointestinal disorders) | 1 (2)
GLUCOSE INTOLERANCE (Metabolism and nutrition disorders) | 1 (2)
HALLUCINATIONS (Psychiatric disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 6 (6)
HEARING IMPAIRED (Ear and labyrinth disorders) | 2 (2)
HEMATURIA (Renal and urinary disorders) | 5 (5)
HEMORRHOIDS (Gastrointestinal disorders) | 1 (1)
HEPATOBILIARY DISORDERS - OTHER, SPECIFY (Hepatobiliary disorders) | 1 (1)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 3 (6)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 1 (2)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 8 (12)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 4 (4)
HYPERKALEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERMAGNESEMIA (Metabolism and nutrition disorders) | 1 (10)
HYPERTENSION (Vascular disorders) | 25 (73)
HYPERURICEMIA (Metabolism and nutrition disorders) | 5 (5)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 9 (30)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 3 (11)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 2 (4)
HYPOKALEMIA (Metabolism and nutrition disorders) | 9 (21)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 6 (8)
HYPONATREMIA (Metabolism and nutrition disorders) | 7 (13)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 4 (15)
HYPOTENSION (Vascular disorders) | 4 (5)
HYPOTHYROIDISM (Endocrine disorders) | 3 (3)
IMMUNE SYSTEM DISORDERS - OTHER, SPECIFY (Immune system disorders) | 2 (2)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 6 (8)
INFUSION RELATED REACTION (General disorders) | 3 (5)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY (Injury, poisoning and procedural complications) | 2 (4)
INR INCREASED (Investigations) | 1 (1)
INSOMNIA (Psychiatric disorders) | 15 (16)
INVESTIGATIONS - OTHER, SPECIFY (Investigations) | 2 (7)
IRON OVERLOAD (Metabolism and nutrition disorders) | 1 (1)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1)
LOCALIZED EDEMA (General disorders) | 1 (1)
LUNG INFECTION (Infections and infestations) | 2 (2)
LYMPHOCYTE COUNT DECREASED (Investigations) | 10 (26)
MEMORY IMPAIRMENT (Nervous system disorders) | 4 (5)
METABOLISM AND NUTRITION DISORDERS - OTHER, SPECIFY (Metabolism and nutrition disorders) | 11 (18)
MUCOSAL INFECTION (Infections and infestations) | 1 (1)
MUCOSITIS ORAL (Gastrointestinal disorders) | 10 (18)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 3 (3)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 5 (8)
MYALGIA (Musculoskeletal and connective tissue disorders) | 4 (6)
NAIL DISCOLORATION (Skin and subcutaneous tissue disorders) | 1 (1)
NAIL RIDGING (Skin and subcutaneous tissue disorders) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 30 (50)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 4 (4)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY (Nervous system disorders) | 4 (5)
NEUTROPHIL COUNT DECREASED (Investigations) | 12 (21)
NON-CARDIAC CHEST PAIN (General disorders) | 3 (3)
OBESITY (Metabolism and nutrition disorders) | 1 (2)
ORAL DYSESTHESIA (Gastrointestinal disorders) | 1 (1)
ORAL PAIN (Gastrointestinal disorders) | 3 (3)
PAIN (General disorders) | 11 (13)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (6)
PALMAR-PLANTAR ERYTHRODYSESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 3 (3)
PALPITATIONS (Cardiac disorders) | 1 (1)
PARESTHESIA (Nervous system disorders) | 3 (7)
PERICARDIAL TAMPONADE (Cardiac disorders) | 1 (1)
PERIORBITAL EDEMA (Skin and subcutaneous tissue disorders) | 1 (2)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 2 (2)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 29 (90)
PHOTOPHOBIA (Eye disorders) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 7 (21)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 1 (1)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (2)
PRURITUS (Skin and subcutaneous tissue disorders) | 3 (5)
PSYCHIATRIC DISORDERS - OTHER, SPECIFY (Psychiatric disorders) | 2 (2)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 2 (3)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 2 (2)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY (Renal and urinary disorders) | 2 (2)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 6 (7)
SINUS TACHYCARDIA (Cardiac disorders) | 2 (2)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 3 (5)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN INFECTION (Infections and infestations) | 1 (1)
SLEEP APNEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 2 (2)
SPASTICITY (Nervous system disorders) | 1 (1)
STOMACH PAIN (Gastrointestinal disorders) | 5 (6)
SYNCOPE (Nervous system disorders) | 4 (4)
THROMBOEMBOLIC EVENT (Vascular disorders) | 7 (7)
TINNITUS (Ear and labyrinth disorders) | 2 (2)
TUMOR LYSIS SYNDROME (Metabolism and nutrition disorders) | 1 (1)
TUMOR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 4 (5)
URINARY FREQUENCY (Renal and urinary disorders) | 2 (3)
URINARY RETENTION (Renal and urinary disorders) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 2 (5)
URINARY TRACT PAIN (Renal and urinary disorders) | 3 (3)
URINARY URGENCY (Renal and urinary disorders) | 3 (3)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1)
VASCULAR DISORDERS - OTHER, SPECIFY (Vascular disorders) | 2 (3)
VERTIGO (Ear and labyrinth disorders) | 2 (4)
VOMITING (Gastrointestinal disorders) | 16 (35)
WEIGHT GAIN (Investigations) | 5 (6)
WEIGHT LOSS (Investigations) | 20 (28)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1)
WHITE BLOOD CELL DECREASED (Investigations) | 9 (23)
WOUND INFECTION (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT03283761/Prot_SAP_000.pdf